CLINICAL TRIAL: NCT03729206
Title: Visualization of Microcirculation in Patients With Leukemic Hyperleukocytosis
Brief Title: Microcirculation in Patients With Leukemic Hyperleukocytosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: leuko_MedA2018
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Hyperleukocytic Syndrome
MeSH Terms: interventions — Intravital Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sublingual microscopy (Experimental)
  Interventions: Diagnostic Test: intravital microscopy

INTERVENTIONS:
Diagnostic Test: intravital microscopy — intravital microscopy with sidestream dark-field imaging

SUMMARY:
Hyperleukocytosis in patients with acute leukemia impacts rheology and microvascularization, leading to severe symptoms or even death. The investigators investigated whether blood stream alterations induced by hyperleukocytosis can be detected by sidestream dark-field imaging and whether they correlate with the grade of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* acute leukemia
* de-novo or relapsed stage
* able to give consent

Exclusion Criteria:

* severe oral mucositis
* unable to give consent
* pregnant women
* patients hospitalized for psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
microvascular flow index (MFI) of sublingual microcirculation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schliemann, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- Universitätsklinikum Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No